CLINICAL TRIAL: NCT02744092
Title: Direct Oral Anticoagulants (DOACs) Versus LMWH +/- Warfarin for VTE in Cancer: A Randomized Effectiveness Trial (CANVAS Trial)
Brief Title: Direct Oral Anticoagulants (DOACs) Versus LMWH +/- Warfarin for VTE in Cancer
Acronym: CANVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-28; CER-1503-29805 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-02

CONDITIONS: Cancer; Venous Thromboembolism; Deep Vein Thrombosis (DVT); Pulmonary Embolism (PE); Blood Clot
Keywords: Rivaroxaban (Xarelto); Apixaban (Eliquis); Edoxaban (Savaysa); Dabigatran (Pradaxa); Warfarin (Coumadin); Low molecular weight heparin (LMWH)
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Thrombosis | interventions — Rivaroxaban; apixaban; edoxaban; Dabigatran; Warfarin; Dalteparin; Enoxaparin; Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Randomized Arm 1 (DOACs) (Active Comparator): Randomized Arm 1 will get anticoagulation therapy with a Direct Oral AntiCoagulant (DOAC). There are four FDA-approved DOAC drugs that may be used for this study: Rivaroxaban, Apixaban, Edoxaban, or Dabigatran. The treatment (including dosage form, dosage, frequency and duration) should be administered in accordance with the drug's FDA package insert, and all modifications are at the discretion of the treating investigator.
  Interventions: Drug: Rivaroxaban; Drug: Apixaban; Drug: Edoxaban; Drug: Dabigatran
- Randomized Arm 2 (LMWH) (Active Comparator): Randomized Arm 2 will get anticoagulation therapy with low molecular weight heparin (LMWH) with or without a transition to warfarin. There are three FDA-approved LMWH drugs that may be used for this study: Dalteparin, Enoxaparin, or Fondaparinux. The treatment (including dosage form, dosage, frequency and duration) should be administered in accordance with the drug's FDA package insert, and all modifications are at the discretion of the treating investigator.
  Interventions: Drug: Warfarin; Drug: Dalteparin; Drug: Enoxaparin; Drug: Fondaparinux
- Preference Cohort 1 (DOACs) (Active Comparator): If an eligible participant is offered randomization and declines randomization, then a limited number of participants (up to N=190) will be allowed to enroll in the Preference Cohort. In this case, the treating physician and patient choose Arm 1 or Arm 2 (non-randomized).
  Preference cohort: Non-randomized Arm 1 will get anticoagulation therapy with a Direct Oral AntiCoagulant (DOAC).
  Interventions: Drug: Rivaroxaban; Drug: Apixaban; Drug: Edoxaban; Drug: Dabigatran
- Preference Cohort 2 (LMWH) (Active Comparator): If an eligible participant is offered randomization and declines randomization, then a limited number of participants (up to N=190) will be allowed to enroll in the Preference Cohort. In this case, the treating physician and patient choose Arm 1 or Arm 2 (non-randomized).
  Preference cohort: Non-randomized Arm 2 will get anticoagulation therapy with Low Molecular Weight Heparin (LMWH) with or without a transition to warfarin.
  Interventions: Drug: Warfarin; Drug: Dalteparin; Drug: Enoxaparin; Drug: Fondaparinux

INTERVENTIONS:
Drug: Rivaroxaban — Anticoagulation therapy.
  Other Names: Xarelto
  Arms: Preference Cohort 1 (DOACs); Randomized Arm 1 (DOACs)
Drug: Apixaban — Anticoagulation therapy.
  Other Names: Eliquis
  Arms: Preference Cohort 1 (DOACs); Randomized Arm 1 (DOACs)
Drug: Edoxaban — Anticoagulation therapy.
  Other Names: Savaysa
  Arms: Preference Cohort 1 (DOACs); Randomized Arm 1 (DOACs)
Drug: Dabigatran — Anticoagulation therapy.
  Other Names: Pradaxa
  Arms: Preference Cohort 1 (DOACs); Randomized Arm 1 (DOACs)
Drug: Warfarin — Anticoagulation therapy.
  Other Names: Coumadin
  Arms: Preference Cohort 2 (LMWH); Randomized Arm 2 (LMWH)
Drug: Dalteparin — Anticoagulation therapy.
  Other Names: Fragmin
  Arms: Preference Cohort 2 (LMWH); Randomized Arm 2 (LMWH)
Drug: Enoxaparin — Anticoagulation therapy.
  Other Names: Lovenox
  Arms: Preference Cohort 2 (LMWH); Randomized Arm 2 (LMWH)
Drug: Fondaparinux — Anticoagulation therapy.
  Other Names: Arixtra
  Arms: Preference Cohort 2 (LMWH); Randomized Arm 2 (LMWH)

SUMMARY:
The overarching objective of the study is to determine the effectiveness of LMWH/ warfarin vs. DOAC anticoagulation for preventing recurrent VTE in cancer patients. The intervention strategy is Direct Oral AntiCoagulants (DOAC) therapy with edoxaban, apixaban, rivaroxaban, or dabigatran. The comparator is low molecular weight heparin (LMWH) alone or with warfarin. The information gained will empower cancer patients and physicians to make more informed choices about anticoagulation strategies to manage VTE.

DETAILED DESCRIPTION:
Venous blood clots affect nearly a million Americans each year. Venous clots in the legs are called deep venous thrombosis (DVT) and are dangerous because they travel to the lungs where they cause blockages known as pulmonary emboli (PE). DVT and PE are called venous thromboemboli (VTE). Cancer is a risk factor with nearly 200,000 VTEs in cancer patients each year. The purpose of VTE treatment is to prevent the initial clot from spreading and to prevent new clots from forming. This is accomplished by thinning the blood, or anticoagulation. Without anticoagulation, VTEs recur and are often fatal.

Recently, the FDA has approved 4 new Direct Oral AntiCoagulants (DOACs) for preventing VTE recurrence. Few cancer patients were included in the efficacy trials, and practice guidelines fall silent on whether switching to DOAC therapy is advisable. To fill this knowledge gap, the Alliance Foundation Trials LLC, a research network of academic and community practices across the US, is conducting a pragmatic randomized effectiveness trial.

The overarching objective of the study is to determine the effectiveness of LMWH/ warfarin vs. DOAC anticoagulation for preventing recurrent VTE in cancer patients. The investigators will conduct a trial of 811 cancer patients followed for 6 months. The intervention strategy is DOAC therapy with edoxaban, apixaban, rivaroxaban, or dabigatran. The comparator is LMWH alone or with warfarin. Within each arm, patients can choose the agent they prefer based on side effects, drug interactions, and practical issues such as co-pays. The trial compares these two strategies in terms of treatment: 1) benefits based on VTE recurrence; 2) harms based on bleeding rates; 3) burdens based on patients' reports of their experiences; and 4) mortality rates.

The investigators hypothesize that the benefits, harms and burdens of DOAC treatment will be non-inferior to, or better than, usual care with LMWH/ warfarin among cancer patients. The information gained will empower cancer patients and physicians to make more informed choices about anticoagulation strategies to manage VTE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced solid tumor cancer, lymphoma, or myeloma (no time restrictions or limitations) -OR- diagnosis of early stage solid tumor cancer, lymphoma, or myeloma <= 12 months prior to study enrollment
* Diagnosis of VTE <= 30 days prior to study enrollment for which potential benefits of anticoagulation therapy to prevent recurrence of VTE are felt by the treating physician to exceed the potential harms

  * Any anticoagulation drug/strategy may be used to treat the index VTE; protocol treatment will begin <= 30days after the index VTE diagnosis date
* Treating physician intends to put participant on anticoagulation therapy for at least three months.
* Age >= 18 years
* Platelet count is >= 50,000/mm^3 (<= 7 days prior to enrollment)
* CrCl (Creatinine Clearance) is >= 15 ml/min (<= 7 days prior to enrollment)

Exclusion Criteria:

* Diagnosis of acute leukemia
* Has ever received or is scheduled to receive an Allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT)

  * Patients who have ever received an Autologous Hematopoietic Stem Cell Transplantation (autoHSCT) ARE eligible.
  * Patients who are scheduled to receive an Autologous Hematopoietic Stem Cell Transplantation (autoHSCT) are NOT eligible
* Ongoing, clinically significant bleeding (CTCAE grade 3 or 4)
* Ongoing therapy with a P-gp inhibitor (e.g., nelfinavir, indinavir, or saquinavir-protease inhibitors for HIV) as these drugs interact with the factor Xa inhibitors
* Therapy with any azole antifungals (e.g., itraconazole, ketaconazole, voriconazole) at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Schrag, MD MPH, Study Chair — Alliance Foundation Trials, LLC.; Jean Connors, MD, Study Chair — Alliance Foundation Trials, LLC.
Locations (151):
- United States (151):
  - South County Hematology, Chula Vista, California
  - Sharp Rees-Stealy, Chula Vista, California
  - Washington Hospital Healthcare System, Fremont, California
  - Washington Hospital, Fremont, California
  - VA Central California Fresno Medical Center, Fresno, California
  - Cancer Center Oncology Medical Group, La Mesa, California
  - Medical Oncology Associates- San Diego, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - UCSF Medical Center - Mission Bay, San Francisco, California
  - Saint Joseph's Medical Center, Stockton, California
  - Middlesex Hospital, Middletown, Connecticut
  - The Stamford Hospital, Stamford, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - Breast Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Hollis Cancer Center, Lakeland, Florida
  - Breast Cancer Center at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - The Center for Cancer Care-Duluth, Duluth, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - The Center for Cancer Care-Snellville, Snellville, Georgia
  - Hawaii Cancer Care POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc Kuakini, Honolulu, Hawaii
  - Kootenai Health, Post Falls, Idaho
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle on Vermillion, Danville, Illinois
  - Carle - Effingham, Effingham, Illinois
  - NorthShore University HealthSystem Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem Highland Park Hospital, Highland Park, Illinois
  - Carle - Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - NorthShore University HealthSystem Skokie ACC, Skokie, Illinois
  - The Carle Foundation Hospital/Carle Cancer Center, Urbana, Illinois
  - Franciscan St. Francis Health - Indianapolis, Indianapolis, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan St. Francis Health - Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital at South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Saint Elizabeth Medical Center Fort Thomas, Fort Thomas, Kentucky
  - Chandler Medical Center - University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Louisville Physicians, PSC, Louisville, Kentucky
  - University of Louisville, Division of Surgical Oncology, Louisville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - DF/BWCC at Milford Regional Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Green Bay Oncology, Ltd./St. Francis Hospital, Escanaba, Michigan
  - Masonic Cancer Center University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Minnesota Health: Clinics and Surgery Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Veterans Administration/Harry S Truman Memorial Hospital, Columbia, Missouri
  - Ellis Fischel Cancer Center University of Missouri Healthcare, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Siteman Cancer Center - West County, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic, Billings, Montana
  - Montana Cancer Consortium, Billings, Montana
  - Bozeman Health, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nevada Cancer Specialists - Oakey, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Nevada Cancer Specialists - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists - Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology PA, Concord, New Hampshire
  - New Hampshire Oncology-Hematology PA, Hooksett, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dana-Farber/New Hampshire Oncology Hematology, Londonderry, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - SUNY Upstate Medical University, New York, New York
  - Mission Hospital - Memorial Campus, Asheville, North Carolina
  - Southeastern Medical Oncology Center, Clinton, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Southeastern Medical Oncology Center, Jacksonville, North Carolina
  - Kenansville Medical Center, Kenansville, North Carolina
  - Kinston Medical Specialists, P.A., Kinston, North Carolina
  - Lenoir Memorial Hospital, Kinston, North Carolina
  - Onslow Medical Center, Richlands, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Dayton Physicians LLC, Miami Valley South, Centerville, Ohio
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Dayton Physicians LLC, Samaritan North, Dayton, Ohio
  - Dayton Clincial Oncology Program, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Wright Patterson Medical Center, Dayton, Ohio
  - Dayton Physicians LLC, Atrium, Franklin, Ohio
  - Dayton Physicians, Wayne, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Toledo Clinic Cancer Center - Maumee, Maumee, Ohio
  - Toledo Clinic Cancer Center - Toledo, Toledo, Ohio
  - Dayton Physicians LLC, Upper valley, Troy, Ohio
  - WellSpan Health Ephrata Cancer Center, Ephrata, Pennsylvania
  - WellSpan Health Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Health Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - WellSpan Health York Cancer Center, York, Pennsylvania
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Augusta Health Cancer Center, Fishersville, Virginia
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Bon Secours Cancer Institute Medical Oncology at Memorial Regional, Mechanicsville, Virginia
  - Bon Secours Cancer Institute Medical Oncology at St. Francis, Midlothian, Virginia
  - Bon Secours Cancer Institute Medical Oncology at St. Mary's, Richmond, Virginia
  - MultiCare Regional Cancer Center - Auburn, Auburn, Washington
  - MultiCare Regional Cancer Center - Gig Harbor Medical Park, Gig Harbor, Washington
  - MultiCare Regional Cancer Center - Puyallup, Puyallup, Washington
  - Multicare Institute for Research & Innovation, Tacoma, Washington
  - MultiCare Regional Cancer Center - Tacoma, Tacoma, Washington
  - Green Bay Oncology, Ltd./HSHS St. Vincent Hospital, Green Bay, Wisconsin
  - HSHS St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Ltd./HSHS St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - HSHS St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Green Bay Oncology, Ltd./HSHS St. Clare Memorial Hospital, Oconto Falls, Wisconsin
  - Green Bay Oncology, Ltd./Door County Memorial Hospital, Sturgeon Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual-level de-identified datasets will be made available to investigators working under an institution with a Federal Wide Assurance (FWA) who formally submit a request to the study chairs at the Dana-Farber Cancer Institute. Prior to the release of datasets, DFCI will ensure certain requirements, e.g., IRB approval and data use agreement, are in place. These datasets will be available within 6 months of publication of the manuscript and following a formal request by an investigator to and approval from DFCI.
Supporting Information: Study Protocol, SAP
Time Frame: within 6 months of publication of the manuscript, no end date
Access Criteria: following a formal request by an investigator to and approval from DFCI

REFERENCES:
- [Derived] Schrag D, Uno H, Rosovsky R, Rutherford C, Sanfilippo K, Villano JL, Drescher M, Jayaram N, Holmes C, Feldman L, Zattra O, Farrar-Muir H, Cronin C, Basch E, Weiss A, Connors JM; CANVAS Investigators. Direct Oral Anticoagulants vs Low-Molecular-Weight Heparin and Recurrent VTE in Patients With Cancer: A Randomized Clinical Trial. JAMA. 2023 Jun 13;329(22):1924-1933. doi: 10.1001/jama.2023.7843. PMID 37266947
- [Derived] Riaz IB, Fuentes HE, Naqvi SAA, He H, Sipra QR, Tafur AJ, Padranos L, Wysokinski WE, Marshall AL, Vandvik PO, Montori V, Bryce AH, Liu H, Badgett RG, Murad MH, McBane RD 2nd. Direct Oral Anticoagulants Compared With Dalteparin for Treatment of Cancer-Associated Thrombosis: A Living, Interactive Systematic Review and Network Meta-analysis. Mayo Clin Proc. 2022 Feb;97(2):308-324. doi: 10.1016/j.mayocp.2020.10.041. Epub 2021 Jun 22. PMID 34172290
- See also: FDA Package Insert for Rivaroxaban (Xarelto) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2011/202439s001lbl.pdf
- See also: FDA Package Insert for Apixaban (Eliquis) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2012/202155s000lbl.pdf
- See also: FDA Package Insert for Edoxaban (Savaysa) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2015/206316lbl.pdf
- See also: FDA Package Insert for Dabigatran (Pradaxa) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2011/022512s007lbl.pdf
- See also: FDA Package Insert for Dalteparin (Fragmin) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/020287s050lbl.pdf
- See also: FDA Package Insert for Enoxaparin (Lovenox) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2009/020164s083lbl.pdf
- See also: FDA Package Insert for Fondaparinux (Arixtra) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/021345s023lbl.pdf
- See also: FDA Package Insert for Warfarin (Coumadin) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2011/009218s107lbl.pdf
- Available data/document: Study Protocol: AFT-28 — https://www.allianceforclinicaltrialsinoncology.org/main/public/standard.xhtml?path=%2FPublic%2FAFT — Email the study team at CANVAS@AllianceFoundationTrials.org.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 67 US-based healthcare institutions between December 2016 and April 2020.
Groups:
- Preference Cohort 1 (DOACs): If an eligible participant is offered randomization and declines randomization, then a limited number of participants (up to N=190) will be allowed to enroll in the Preference Cohort. In this case, the treating physician and patient choose Arm 1 or Arm 2 (non-randomized).
  Preference cohort: Non-randomized Arm 1 will get anticoagulation therapy with a Direct Oral AntiCoagulant (DOAC).
  Rivaroxaban: Anticoagulation therapy.
  Apixaban: Anticoagulation therapy.
  Edoxaban: Anticoagulation therapy.
  Dabigatran: Anticoagulation therapy.
- Preference Cohort 2 (LMWH): If an eligible participant is offered randomization and declines randomization, then a limited number of participants (up to N=190) will be allowed to enroll in the Preference Cohort. In this case, the treating physician and patient choose Arm 1 or Arm 2 (non-randomized).
  Preference cohort: Non-randomized Arm 2 will get anticoagulation therapy with Low Molecular Weight Heparin (LMWH) with or without a transition to warfarin.
  Dalteparin: Anticoagulation therapy.
  Enoxaparin: Anticoagulation therapy.
  Fondaparinux: Anticoagulation therapy.
Period: Enrolled & Received Selected Treatment
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Started | 335 | 336 | 108 | 32
Received Assigned Treatment (Apixaban) | 193 | 0 | 57 | 0
Received Assigned Treatment (Rivaroxaban) | 122 | 0 | 48 | 0
Received Assigned Treatment (Dabigatran) | 9 | 0 | 2 | 0
Received Assigned Treatment (Edoxaban) | 6 | 0 | 0 | 0
Received Assigned Treatment (Enoxaparin) | 0 | 277 | 0 | 24
Received Assigned Treatment (Fondaparinux) | 0 | 23 | 0 | 6
Received Assigned Treatment (Dalteparin) | 0 | 8 | 0 | 0
Did Not Receive Assigned/Selected Treatment | 5 | 28 | 1 | 2
Completed | 330 | 308 | 107 | 30
Not Completed | 5 | 28 | 1 | 2
Period: 6-Month Clinical Outcomes(Chart Review)
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Started | 330 | 308 | 107 | 30
Completed | 330 | 308 | 107 | 30
Not Completed | 0 | 0 | 0 | 0
Period: 3-Month Patient-Reported Outcomes Survey
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Started | 330 | 308 | 107 | 30
Approached for 3-month Survey | 295 | 280 | 99 | 26
Completed | 212 | 197 | 77 | 16
Not Completed | 118 | 111 | 30 | 14
Period: 6-Month Patient-Reported Outcomes Survey
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Started (All patients were eligible to be included in the 6-month survey, regardless of whether or not they completed the 3-month survey.) | 330 | 308 | 107 | 30
Approached for 6-month Survey | 262 | 253 | 89 | 21
Completed | 191 | 177 | 75 | 12
Not Completed | 139 | 131 | 32 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH) | Total
Number analyzed (Participants) | 330 | 308 | 107 | 30 | 775
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 175 | 197 | 45 | 11 | 428
  >=65 years | 155 | 111 | 62 | 19 | 347
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age, median (q1, q3) | 64 [56 to 70] | 62 [54 to 68] | 66 [58 to 72] | 67 [61 to 72] | 64 [55 to 70]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 181 | 172 | 51 | 18 | 422
  Male | 149 | 136 | 56 | 12 | 353
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 3 | 0 | 33
  Not Hispanic or Latino | 306 | 287 | 101 | 28 | 722
  Unknown or Not Reported | 9 | 6 | 3 | 2 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 1 | 1 | 5
  Asian | 4 | 6 | 2 | 2 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 2
  Black or African American | 39 | 38 | 12 | 3 | 92
  White | 277 | 255 | 90 | 23 | 645
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 8 | 2 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Non-Fatal VTE Recurrence at 6 Months (%)
Description: To compare the effectiveness of anticoagulation with a DOAC (intervention) with LMWH/warfarin (comparator) for preventing VTE recurrence in patients with cancer based on cumulative VTE recurrence reported by patients or clinicians at 6 months. Only VTEs that were nonfatal were considered because of the challenges of attributing cause of death in cancer patients to tumor progression vs. VTE.
Time Frame: 6 months
Population: Primary analyses were performed on the participants who began protocol-directed therapy, the "as treated" population.
Measure: Number; unit: percentage of patients
Groups:
- Preference Cohort 2 (LMWH): If an eligible participant is offered randomization and declines randomization, then a limited number of participants (up to N=190) will be allowed to enroll in the Preference Cohort. In this case, the treating physician and patient choose Arm 1 or Arm 2 (non-randomized).
  Preference cohort: Non-randomized Arm 2 will get anticoagulation therapy with Low Molecular Weight Heparin (LMWH) with or without a transition to warfarin.
  Warfarin: Anticoagulation therapy.
  Dalteparin: Anticoagulation therapy.
  Enoxaparin: Anticoagulation therapy.
  Fondaparinux: Anticoagulation therapy.
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 330 | 308 | 107 | 30
percentage of patients | 6.1 | 8.8 | 7.5 | 4.1

2. Secondary Outcome: Cumulative Rates of Major Bleeding
Description: To compare the harms of DOAC vs. LMWH/warfarin therapy for cancer patients with VTE based on the cumulative rate of major bleeding at 6 months. d. Major bleeding was defined as Grade >=3 on the Common Terminology Criteria for Adverse Events from the National Cancer Institute (NCI CTCAE) criteria version 5.0 (i.e., severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living).
Time Frame: 6 months
Population: Primary analyses were performed on the participants who began protocol-directed therapy, the "as treated" population.
Measure: Number; unit: percentage of patients
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 330 | 308 | 107 | 30
percentage of patients | 5.2 | 5.6 | 11.5 | 7.6

3. Secondary Outcome: Health Related Quality of Life Reported by Participants Via the Optum SF-12v2 Health Survey Questionnaire
Description: Change in physical health at 3 months. Health-related quality of life was measured using the 12-Item Short Form Health Survey (SF-12) sub-scales for physical and mental health (score range, 0-100; higher scores indicate better physical and mental health functioning). Survey content included minor verbiage changes for clarity. The presented scores in this results section indicate the change (difference) in mean scores between the baseline and 3-month follow-up assessment.
Time Frame: 3 months
Population: Participants completing the 3-month survey assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 212 | 197 | 77 | 16
units on a scale | 1.8 [0.6 to 3.0] | 0.7 [-0.5 to 2.0] | 3.4 [0.4 to 6.3] | -0.3 [-8.7 to 8.1]

4. Secondary Outcome: Burden of Anticoagulation Therapy Reported by Participants Via the Anti-Clot Treatment Scale (ACTS) Questionnaire
Description: To compare the burden of anticoagulation therapy with DOAC vs. with LMWH/warfarin for cancer patients with VTE at 3 months. The burden scale has12 items and patients are asked to rate their experiences on a 5-point scale of intensity (1=not at all, 2=a little, 3=moderately, 4=quite a bit, 5=extremely). The ACTS burden tool is then scored using the totals from each question with a total score from 12 to 60 possible. Higher scores signify greater satisfaction (lower burden).
Time Frame: 3 months
Population: Participants completing the 3-month survey assessment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 212 | 197 | 77 | 16
score on a scale | 56.7 [56.1 to 57.3] | 53.3 [52.5 to 54.2] | 55.8 [54.8 to 56.9] | 54.9 [52.4 to 57.4]

5. Secondary Outcome: Mortality Reported by Participants' Surrogates (Via Study-specific Questionnaire) or Clinicians (Via Study-specific Case Report Form)
Description: To compare the impact of DOAC vs. LMWH/warfarin therapy on mortality in cancer patients with VTE based on survival at 6 months. Mortality was reported by participants' surrogates (via study-specific questionnaire) or clinicians (via study-specific case report form)
Time Frame: 6 months
Population: Primary analyses were performed on the participants who began protocol-directed therapy, the "as treated" population.
Measure: Number; unit: percentage of patients
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 330 | 308 | 107 | 30
percentage of patients | 21.5 | 18.4 | 16.3 | 23.8

6. Secondary Outcome: Health Related Quality of Life Reported by Participants Via the Optum SF-12v2 Health Survey Questionnaire
Description: Change in physical health at 6 months. Health-related quality of life was measured using the 12-Item Short Form Health Survey (SF-12) sub-scales for physical and mental health (score range, 0-100; higher scores indicate better physical and mental health functioning). Survey content included minor verbiage changes for clarity. The presented scores in this results section indicate the change (difference) in mean scores between the baseline and 6-month follow-up assessment.
Time Frame: 6 months
Population: Participants completing the 6-month survey assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 191 | 177 | 75 | 12
units on a scale | 2.4 [0.9 to 3.8] | 0.7 [-0.8 to 2.2] | 2.1 [-0.3 to 4.5] | -2.8 [-10.4 to 4.9]

7. Secondary Outcome: Burden of Anticoagulation Therapy Reported by Participants Via the Anti-Clot Treatment Scale (ACTS) Questionnaire
Description: To compare the burden of anticoagulation therapy with DOAC vs. with LMWH/warfarin for cancer patients with VTE at 6 months. The burden scale has12 items and patients are asked to rate their experiences on a 5-point scale of intensity (1=not at all, 2=a little, 3=moderately, 4=quite a bit, 5=extremely). The ACTS burden tool is then scored using the totals from each question with a total score from 12 to 60 possible. Higher scores signify greater satisfaction (lower burden).
Time Frame: 6 months
Population: Participants completing the 6-month survey assessment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 191 | 177 | 75 | 12
score on a scale | 56.5 [55.8 to 57.1] | 54.1 [53.2 to 55.1] | 54.9 [53.4 to 56.4] | 53.1 [49.8 to 56.3]

8. Secondary Outcome: Benefit of Anticoagulation Therapy Reported by Participants Via the Anti-Clot Treatment Scale (ACTS) Questionnaire
Description: To compare the benefit of anticoagulation therapy with DOAC vs. with LMWH/warfarin for cancer patients with VTE at 3 months. The benefits scale has 3 items and patients are asked to rate their experiences on a 5-point scale of intensity (1=not at all, 2=a little, 3=moderately, 4=quite a bit, 5=extremely). The ACTS benefits tool is then scored using the totals from each question with a total score from 3 to 15 possible. Higher scores signify greater satisfaction (greater benefits).
Time Frame: 3-months
Population: Participants completing the 3-month survey assessment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 212 | 197 | 77 | 16
score on a scale | 11.2 [10.7 to 11.6] | 10.7 [10.3 to 11.2] | 10.3 [9.6 to 11.0] | 10.5 [8.9 to 12.1]

9. Secondary Outcome: Benefit of Anticoagulation Therapy Reported by Participants Via the Anti-Clot Treatment Scale (ACTS) Questionnaire
Description: To compare the benefit of anticoagulation therapy with DOAC vs. with LMWH/warfarin for cancer patients with VTE at 6 months. The benefits scale has 3 items and patients are asked to rate their experiences on a 5-point scale of intensity (1=not at all, 2=a little, 3=moderately, 4=quite a bit, 5=extremely). The ACTS benefits tool is then scored using the totals from each question with a total score from 3 to 15 possible. Higher scores signify greater satisfaction (greater benefits).
Time Frame: 6-months
Population: Participants completing the 6-moth survey assessment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 191 | 177 | 75 | 12
score on a scale | 11.6 [11.1 to 12.1] | 11.3 [10.8 to 11.8] | 11.5 [10.8 to 12.1] | 10.1 [8.6 to 11.6]

10. Secondary Outcome: Health Related Quality of Life (Mental Health) Reported by Participants Via the Optum SF-12v2 Health Survey Questionnaire at 3-months
Description: Change in mental health at 3 months from baseline. Health-related quality of life was measured using the 12-Item Short Form Health Survey (SF-12) sub-scales for physical and mental health (score range, 0-100; higher scores indicate better physical and mental health functioning). Survey content included minor verbiage changes for clarity. The scores indicate change in score from baseline.
Time Frame: 3-months
Population: Participants completing the 3-month survey assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 212 | 197 | 77 | 16
units on a scale | -0.3 [-1.8 to 1.1] | 0.7 [-0.6 to 2.1] | 0.3 [-2.1 to 2.6] | 0.4 [-4.5 to 5.3]

11. Secondary Outcome: Health Related Quality of Life (Mental Health) Reported by Participants Via the Optum SF-12v2 Health Survey Questionnaire at 6-months
Description: Change in mental health at 6 months from baseline. Health-related quality of life was measured using the 12-Item Short Form Health Survey (SF-12) sub-scales for physical and mental health (score range, 0-100; higher scores indicate better physical and mental health functioning). Survey content included minor verbiage changes for clarity. The scores indicate change in score from baseline.
Time Frame: 6-months
Population: Participants completing the 6-month survey assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
Number analyzed (Participants) | 191 | 177 | 75 | 12
units on a scale | 0.3 [-1.1 to 1.7] | 0.9 [-0.5 to 2.3] | 1.1 [-1.1 to 3.3] | -1.9 [-7.0 to 3.3]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected for 6-months.
Description: AEs were reported by physicians. Grade 3+ AEs were severe. Other AEs are grade 1 or 2 . Other AE section reports on events that were experienced in >1% of patients, so total # of patients may not match the # of patients experiencing events. We did not report AEs by individual drug arm because we did not randomize drugs; comparisons amongst drugs will be subject to selection bias. Also, the protocol allowed patients to switch drugs, so it would be unclear which AE is affiliated with which drug.
Arm/Group | Randomized Arm 1 (DOACs) | Randomized Arm 2 (LMWH) | Preference Cohort 1 (DOACs) | Preference Cohort 2 (LMWH)
All-Cause Mortality (participants affected / at risk) | 70/330 | 56/308 | 18/107 | 9/30
Serious Adverse Events (participants affected / at risk) | 123/330 | 114/308 | 51/107 | 16/30
Other Adverse Events (participants affected / at risk) | 6/330 | 11/308 | 3/107 | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Arm 1 (DOACs) (N=330) | Randomized Arm 2 (LMWH) (N=308) | Preference Cohort 1 (DOACs) (N=107) | Preference Cohort 2 (LMWH) (N=30)
Anemia (Blood and lymphatic system disorders) | 15 | 10 | 7 | 3 — Grade 3+
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 — Grade 3+
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 — Grade 3+
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2 | 0 — Grade 3+
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 — Grade 3+
Cardiac arrest (Cardiac disorders) | 3 | 2 | 0 | 0 — Grade 3+
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0 | 0 — Grade 3+
Heart failure (Cardiac disorders) | 1 | 2 | 0 | 0 — Grade 3+
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 — Grade 3+
Pericardial tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 — Grade 3+
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 — Grade 3+
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 1 | 0 — Grade 3+
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 — Grade 3+
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 0 | 0 — Grade 3+
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0 — Grade 3+
Colitis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 — Grade 3+
Colonic obstruction (Gastrointestinal disorders) | 3 | 0 | 0 | 0 — Grade 3+
Colonic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Grade 3+
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 0 | 1 — Grade 3+
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 — Grade 3+
Esophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 — Grade 3+
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Grade 3+
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Grade 3+
Lower GI hemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 0 — Grade 3+
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Grade 3+
Nausea (Gastrointestinal disorders) | 3 | 4 | 1 | 1 — Grade 3+
Obstruction gastric (Gastrointestinal disorders) | 1 | 1 | 1 | 0 — Grade 3+
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Grade 3+
Rectal hemorrhage (Gastrointestinal disorders) | 4 | 3 | 2 | 0 — Grade 3+
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Grade 3+
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 1 | 1 — Grade 3+
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 2 | 1 | 0 — Grade 3+
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0 | 0 — Grade 3+
Abdominal pain (Gastrointestinal disorders) | 8 | 3 | 3 | 3 — Grade 3+
Death NOS (General disorders) | 34 | 33 | 5 | 1 — Grade 3+
Edema limbs (General disorders) | 2 | 0 | 0 | 1 — Grade 3+
Fatigue (General disorders) | 4 | 1 | 3 | 0 — Grade 3+
Fever (General disorders) | 1 | 1 | 0 | 0 — Grade 3+
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0 — Grade 3+
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 0 — Grade 3+
Pain (General disorders) | 1 | 4 | 0 | 1 — Grade 3+
Sudden death NOS (General disorders) | 2 | 0 | 0 | 1 — Grade 3+
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 | 0 | 0 — Grade 3+
Generalized edema (General disorders) | 0 | 1 | 0 | 0 — Grade 3+
Disease progression (General disorders) | 22 | 7 | 2 | 0 — Grade 3+
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0 | 1 — Grade 3+
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1 | 1 | 0 — Grade 3+
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0 — Grade 3+
Abdominal infection (Infections and infestations) | 1 | 0 | 1 | 0 — Grade 3+
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 — Grade 3+
Breast infection (Infections and infestations) | 0 | 1 | 0 | 0 — Grade 3+
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 1 | 0 — Grade 3+
Joint infection (Infections and infestations) | 0 | 0 | 0 | 1 — Grade 3+
Lung infection (Infections and infestations) | 6 | 5 | 6 | 1 — Grade 3+
Peritoneal infection (Infections and infestations) | 0 | 1 | 0 | 0 — Grade 3+
Sepsis (Infections and infestations) | 3 | 5 | 2 | 2 — Grade 3+
Skin infection (Infections and infestations) | 1 | 1 | 0 | 0 — Grade 3+
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 | 0 — Grade 3+
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 3 | 0 — Grade 3+
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 4 | 1 — Grade 3+
Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 — Grade 3+
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 — Grade 3+
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 — Grade 3+
Blood bilirubin increased (Investigations) | 2 | 1 | 0 | 0 — Grade 3+
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0 | 0 — Grade 3+
GGT increased (Investigations) | 0 | 0 | 1 | 0 — Grade 3+
INR incresed (Investigations) | 0 | 1 | 0 | 0 — Grade 3+
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0 — Grade 3+
Neutrophil count decreased (Investigations) | 1 | 1 | 2 | 0 — Grade 3+
Platelet count decreased (Investigations) | 3 | 5 | 1 | 0 — Grade 3+
White blood cell decreased (Investigations) | 0 | 1 | 1 | 0 — Grade 3+
Dehydration (Metabolism and nutrition disorders) | 6 | 1 | 1 | 1 — Grade 3+
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 — Grade 3+
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 — Grade 3+
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 — Grade 3+
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 — Grade 3+
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — Grade 3+
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 — Grade 3+
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 — Grade 3+
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 — Grade 3+
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 — Grade 3+
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — Grade 3+
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 — Grade 3+
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — Grade 3+
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 13 | 12 | 5 — Grade 3+
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 — Grade 3+
Cognitive disturbance (Nervous system disorders) | 1 | 1 | 0 | 0 — Grade 3+
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 — Grade 3+
Edema cerebral (Nervous system disorders) | 0 | 1 | 0 | 0 — Grade 3+
Facial muscle weakness (Nervous system disorders) | 0 | 1 | 0 | 0 — Grade 3+
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 — Grade 3+
Hydrocephalus (Nervous system disorders) | 2 | 0 | 0 | 0 — Grade 3+
Intracranial hemorrhage (Nervous system disorders) | 1 | 2 | 1 | 0 — Grade 3+
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0 | 0 | 0 — Grade 3+
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 — Grade 3+
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 — Grade 3+
Stroke (Nervous system disorders) | 5 | 1 | 0 | 0 — Grade 3+
Syncope (Nervous system disorders) | 0 | 0 | 4 | 0 — Grade 3+
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 — Grade 3+
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 — Grade 3+
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 — Grade 3+
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 — Grade 3+
Acute kidney injury (Renal and urinary disorders) | 3 | 3 | 1 | 0 — Grade 3+
Hematuria (Renal and urinary disorders) | 4 | 2 | 1 | 2 — Grade 3+
Urinary tract obstruction (Renal and urinary disorders) | 1 | 2 | 0 | 0 — Grade 3+
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 0 | 1 | 0 — Grade 3+
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 — Grade 3+
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 — Grade 3+
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 — Grade 3+
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Grade 3+
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — Grade 3+
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 — Grade 3+
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1 | 2 — Grade 3+
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 — Grade 3+
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 0 — Grade 3+
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 — Grade 3+
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Grade 3+
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 3 | 1 — Grade 3+
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 — Grade 3+
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 — Grade 3+
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 — Grade 3+
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Grade 3+
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 | 1 | 0 | 0 — Grade 3+
Hematoma (Vascular disorders) | 0 | 4 | 0 | 0 — Grade 3+
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 — Grade 3+
Hypotension (Vascular disorders) | 1 | 1 | 1 | 1 — Grade 3+
Thromboembolic event (Vascular disorders) | 14 | 16 | 5 | 1 — Grade 3+
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 0 | 0 — Grade 3+
Arterial thromboembolism (Vascular disorders) | 1 | 0 | 0 | 0 — Grade 3+
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Arm 1 (DOACs) (N=330) | Randomized Arm 2 (LMWH) (N=308) | Preference Cohort 1 (DOACs) (N=107) | Preference Cohort 2 (LMWH) (N=30)
Hematoma (Vascular disorders) | 0 | 2 | 0 | 2 — Grade 1 or 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 — Grade 1 or 2
Anemia (Blood and lymphatic system disorders) | 0 | 5 | 1 | 0 — Grade 1 or 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — Grade 1 or 2
Blurred vision (Eye disorders) | 0 | 0 | 0 | 1 — Grade 1 or 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Grade 1 or 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Grade 1 or 2
Nausea (Gastrointestinal disorders) | 3 | 0 | 2 | 0 — Grade 1 or 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0 — Grade 1 or 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 4 | 1 | 1 — Grade 1 or 2
Fever (General disorders) | 5 | 2 | 3 | 1 — Grade 1 or 2
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — Grade 1 or 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 — Grade 1 or 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 — Grade 1 or 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 — Grade 1 or 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 — Grade 1 or 2
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0 — Grade 1 or 2
Stroke (Nervous system disorders) | 0 | 0 | 1 | 1 — Grade 1 or 2
Confusion (Psychiatric disorders) | 1 | 1 | 0 | 1 — Grade 1 or 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 1 — Grade 1 or 2
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 — Grade 1 or 2
Thromboembolic event (Vascular disorders) | 5 | 11 | 2 | 1 — Grade 1 or 2

LIMITATIONS AND CAVEATS:
This study has several limitations. First, participants and physicians were not blinded to treatment assignment. Second, because participants were randomized within 30 days of a new VTE diagnosis, some were treated with different therapy before randomization. Third, in patients with advanced-stage cancer, it was not possible to distinguish VTE from cancer as the cause of death. Fourth, the included population limits generalizability. Fifth, detailed medication diaries were not obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Complete study results are available in JAMA.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT02744092/Prot_SAP_000.pdf